CLINICAL TRIAL: NCT07387627
Title: Effectiveness of the Coping With and Caring for Infants With Special Needs Program in Infants at Risk of Neurodevelopmental Disorders. A Comparison With Conventional Pediatric Physiotherapy Models and Parent Training
Brief Title: Effectiveness of the COPCA Program in Infants at Risk of Neurodevelopmental Disorders
Acronym: COPCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, PT, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SICEIA-2025-003712; SICEIA-2025-003712 (Registry Identifier: COPCA.01)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neurodevelopmental Disorders; Neurodevelopmental Disorders and Developmental Abnormalities
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- In-person COPCA® Intervention (Experimental): COPCA®-based intervention focused on caregiver coaching and promotion of infant motor initiative and variability. One weekly in-person session at the family home, up to 45 minutes, for 6 months.
  Interventions: Other: Coping with and Caring for Infants with Special Needs
- Online COPCA® Intervention (Active Comparator): COPCA®-based intervention delivered via videoconferencing, focused on caregiver coaching and infant motor initiative and variability. One weekly session of up to 45 minutes for 6 months, following an initial in-person assessment.
  Interventions: Other: Parental Education Program
- Parental Education Group (Active Comparator): Online group-based parental education on motor development and home stimulation, without individualized child intervention. Sessions of 90 minutes every two weeks for 6 months.
  Interventions: Other: Conventional Pediatric Physiotherapy
- Conventional Pediatric Physiotherapy (Active Comparator): Standard pediatric physiotherapy delivered according to usual clinical practice in Early Intervention services, with therapist-led sessions using structured exercises and movement facilitation techniques.
  Interventions: Other: Coping with and Caring for Infants with Special Needs

INTERVENTIONS:
Other: Coping with and Caring for Infants with Special Needs — COPCA®-based intervention focused on caregiver coaching and promotion of infant motor initiative and variability. Delivered weekly for up to 45 minutes over 6 months, either in person or online after an initial in-person assessment, integrated into daily routines and emphasizing self-exploration.
  Arms: Conventional Pediatric Physiotherapy; In-person COPCA® Intervention
Other: Parental Education Program — Online group-based parental education on motor development and home stimulation, delivered in 90-minute sessions every two weeks for 6 months, without individualized child intervention.
  Arms: Online COPCA® Intervention
Other: Conventional Pediatric Physiotherapy — Standard pediatric physiotherapy delivered according to routine clinical practice in Early Intervention services. The intervention consists of therapist-led sessions using structured exercises and movement facilitation techniques, with frequency and duration determined by the reference center.
  Arms: Parental Education Group

SUMMARY:
The purpose of this clinical trial is to evaluate whether the COPCA® program (Coping with and Caring for Infants with Special Needs) is more effective than conventional pediatric physiotherapy and parent education in improving development in infants at risk of neurodevelopmental disorders, as well as empowering their families.

This study will include infants younger than 12 months of corrected age who are at risk of neurodevelopmental disorders and are currently receiving early intervention or pediatric physiotherapy services, together with their parents or primary caregivers.

The main questions this study aims to answer are:

Does the COPCA® program improve motor development and functional abilities in infants at risk of neurodevelopmental disorders more than conventional pediatric physiotherapy or parent education?

Does the COPCA® program increase family empowerment and improve parents' perception of the care they receive compared with traditional intervention models?

The researchers will compare outcomes across four study groups:

In-person COPCA® intervention

Online COPCA® intervention

Parent education group

Conventional pediatric physiotherapy group

Participants will be randomly assigned to one of the four groups. The intervention period will last 6 months, with assessments conducted at the start of the study, during the intervention, and during follow-up.

Infants will take part in age-appropriate daily activities and play situations. Parents or caregivers will actively participate in the intervention sessions and will be supported in learning how to promote their child's development during everyday routines.

The study will assess infant motor development, functional abilities, overall development, family empowerment, and parents' perception of family-centered care using validated assessment tools and interviews. The results of this study may help improve early intervention strategies for infants at risk of neurodevelopmental disorders and support more family-centered approaches to care.

ELIGIBILITY:
Inclusion Criteria:

* Infants at risk of neurodevelopmental disorders.
* Participation in pediatric physiotherapy and/or Early Intervention programs at the time of study inclusion, regardless of the reference center.
* Corrected age under 12 months at the time of recruitment.

Exclusion Criteria:

* Infants with confirmed neurodevelopmental disorders at the time of inclusion.
* Presence of additional medical conditions requiring complex medical or surgical interventions that could interfere with participation in the study (e.g., recent or planned surgery).
* Severe family socio-communicative difficulties that limit participation in coaching sessions (e.g., significant language barriers).

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Infant Motor Profile (IMP) | Baseline, during intervention (3 months), post-intervention (6 months) and follow up (3 and 6 months after intervention)
  Assessment of motor development and quality of motor behavior in infants. The IMP total score ranges from 0 to 100, where higher scores indicate better motor performance and motor behavior quality.
Pediatric Evaluation of Disability Inventory (PEDI) | Baseline, during intervention (3 months), post-intervention (6 months) and follow-up after intervention (3 and 6 months)
  Assessment of functional abilities and performance in daily activities. Scaled scores range from 0 to 100, where higher scores indicate better functional performance and greater independence.
Merrill-Palmer-Revised Scales of Development (MP-R) | Baseline, post-intervention (6 months) and follow-up (6 months after intervention)
  Assessment of overall development across cognitive, motor, and socio-emotional domains. Higher scores indicate higher developmental functioning. The score varies according to age so it does not have a general fixed minimum or maximum value.
Measurement of Processes of Care (MPOC-20) | Post-intervention (6 months)
  Assessment of caregivers' perception of family-centered care. Items are rated on a 7-point Likert scale (1 to 7), where higher scores indicate a higher perception of family-centered care.

SECONDARY OUTCOMES:
Family Empowerment Scale (FES) | Post-intervention (6 months)
  Assessment of family empowerment and perceived impact of the intervention. Items are rated on a 5-point Likert scale (1 to 5), where higher scores indicate greater family empowerment.
Semi-structured interview | Post-intervention (6 months)
  Qualitative exploration of family experiences, perceived usefulness of the intervention, and challenges in home implementation. This outcome does not use a numerical scale. Data will be analyzed using qualitative content analysis.

IPD SHARING:
Plan to Share IPD: Yes
Sharing data
Supporting Information: Study Protocol
Time Frame: For a year since the study ends